CLINICAL TRIAL: NCT01928459
Title: A Phase Ib, Open-label Study of Oral BGJ398 in Combination With Oral BYL719 in Adult Patients With Select Advanced Solid Tumors
Brief Title: Phase 1b Trial of BGJ398/BYL719 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398X2102
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2017-08

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: BGJ398; BYL719; advanced solid tumor; metastatic breast cancer; PK3CA; FGFR; fibroblast growth factor receptor
MeSH Terms: conditions — Breast Neoplasms; Acrocephalosyndactylia | interventions — infigratinib; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metastatic breast cancer (Experimental): Evaluation of safety and efficacy in patients with metastatic breast cancer whose tumors contain mutations to PIK3CA and alterations FGFR 1-3.
  Interventions: Drug: BGJ398; Drug: BYL719
- Solid tumor arm 1 (Experimental): Patients with solid tumors (except for colorectal cancer) whose tumors express mutations to PIK3CA.
  Interventions: Drug: BGJ398; Drug: BYL719
- Solid tumor arm 2 (Experimental): Patients with solid tumors (except for colorectal cancer) whose tumomrs express mutations to PIK3CA and alterations to FGFR 1-3
  Interventions: Drug: BGJ398; Drug: BYL719
- Dose escalation (Experimental): To determine the MTD or RDE of the combination of BGJ398 with BYL719 in patients with advanced or metastastic solid tumors that express mutations to PIK3CA.
  Interventions: Drug: BGJ398; Drug: BYL719

INTERVENTIONS:
Drug: BGJ398 — BGJ398 will be administered orally once daily for the first 21 days of each 28-day cycle.
Drug: BYL719 — BYL719 will be administered orally once daily on each day of the 28-day cycle.

SUMMARY:
To study the safety and efficacy of the combination of BGJ398 with BYL719 in patients whose tumors express mutations to PIK3CA with or without alterations to FGFR 1-3.

DETAILED DESCRIPTION:
This dose escalation/dose expansion study will evaluate the combination of orally administered BGJ398 in combination with orally administered BYL719. During the dose escalation part, the MTD of the combination will be determined in patients whose advanced or metastatic tumors express mutations to PIK3CA. Once the MTD has been determined, the expansion part will begin. Patients will be addd to one of three arms based on the disease type and genetic changes. Patients with metastatic colorectal cancer are not eligible for participation in the expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed advanced or metastatic solid tumors who have failed standard therapy or for whom no effective standard anti-cancer therapy exists
* Documented PIK3CA mutations in all patients in dose escalation and expansion with or without documented genetic alterations in FGFR depending upon dose expansion cohort (either local or central determination)
* Measurable disease defined by RECIST v1.1
* ECOG performance status of ≤2

Exclusion Criteria:

* Prior PI3Ki or selective FGFR inhibitor treatment (for patients enrolled to expansion part)
* Colorectal cancer (for patients enrolled to expansion part)
* Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with fasting glucose ≥ 140 mg/dL / 7.8 mmol/L, history of clinically significant gestational diabetes mellitus or documented steroid-induced diabetes mellitus
* Use of medications that increase serum levels of phosphorus and/or calcium
* Inorganic phosphorus outside of normal limits
* Total and ionized serum calcium outside of normal limits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) of the combination of BGJ398 with BYL719 | Approximately 8 months
  The dose escalation part of the study will be guided by a well-established statistical method/model to estimate the maximum tolerated dose(s) and/or the recommended dose for expansion (RDE). Safety(incidence and nature of DLTs), pharmacokinetic and pharmacodynamic data will guide dose escalation decisioins.

SECONDARY OUTCOMES:
Safety and tolerability of BGJ398/BYL719 combination at the recommended dose for expansion (RDE) | Every 28 days from baseline visit until end of study visit
  This will be assessed by looking at the number of Adverse Events (AEs), serious AEs (SAEs) changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions and reductions
Overall response rate | Every two months from the date of baseline CT scan
  Assessment of preliminary antitumor activity of the combination of BGJ398 with BYL719; Overall response rate = complete response + partial response
Progression free survival | Every two months from the date of baseline CT scan
  Assessment of preliminary antitumor activity of the combination of BGJ398 with BYL719
Time vs. concentration profile of BGJ398 and BYL719 | Every 28 days for up to 10 cycles
  Plasma concentration versus time profiles. Plasma PK parameters will be used to characterize the PK profiles of the combination of BGJ398 with BYL719

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (7):
  - H. Lee Moffitt Cancer Center & Research Institute Moffitt 4, Tampa, Florida
  - University of Michigan Comprehensive Cancer Center SC, Ann Arbor, Michigan
  - Karmanos Cancer Institute Dept of Onc, Detroit, Michigan
  - Washington University School of Medicine Onc Dept, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Onc Dept, New York, New York
  - Vanderbilt University Medical Center Dept of Onc, Nashville, Tennessee
  - Cancer Therapy & Research Center / UT Health Science Center SC, San Antonio, Texas
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Saint-Herblain
- Novartis Investigative Site, Cologne, North Rhine-Westphalia, Germany
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CBGJ398X2102 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16593